CLINICAL TRIAL: NCT06293469
Title: Accelerated Flap Coverage Versus Standard Timing in the Treatment of Severe Lower Extremity Musculoskeletal Injuries
Brief Title: Accelerated Flap Coverage in Severe Lower Extremity Trauma
Acronym: FLAP ATTACK
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: McMaster University (Other); University of Maryland, Baltimore (Other); Orthopaedic Trauma Association (Other); Foundation of Orthopedic Trauma (Other); National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH); Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB00434587
Record Dates: First submitted 2024-02-28; First posted 2024-03-05 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-10

CONDITIONS: Open Tibia Fracture; Open Dislocation of Ankle; Extremity Fracture Lower; Extremity Injuries Lower
MeSH Terms: conditions — Leg Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Accelerated Flap Coverage (Experimental): Accelerated flap surgery timing at a goal of within 72 hours from injury. Management of the fracture or dislocation, selection of flap, and post-injury flap management will be at the discretion of the operating surgeons and documented for both treatment groups.
  Interventions: Procedure: Accelerated Flap Coverage Surgery
- Standard of Care Flap Timing (Active Comparator): The flap surgery will be performed at the standard of care timing for the institution. Management of the fracture or dislocation, selection of flap, and post-injury flap management will be at the discretion of the operating surgeons and documented for both treatment groups.
  Interventions: Procedure: Standard of Care Flap Timing

INTERVENTIONS:
Procedure: Accelerated Flap Coverage Surgery — Timing of the flap surgery is with a goal of 72 hours from injury
  Arms: Accelerated Flap Coverage
Procedure: Standard of Care Flap Timing — Timing of the flap surgery is the standard of care flap timing for the participating institution.
  Arms: Standard of Care Flap Timing

SUMMARY:
The goal of this randomized controlled trial is to determine if accelerated flap coverage compared to standard flap coverage timing leads to improved infection-related complications in patients with open fractures and/or dislocations below the knee. Eligible patients will be randomized to receive either a flap within a goal of 72 hours of injury or standard of care flap timing for the institution. The primary outcome will be a composite outcome to evaluate clinical status 6 months after randomization. Components of the composite outcome will be hierarchically assessed in the following order: 1) all-cause mortality, 2) amputation related to injury, 3) re-operation for infection and/or flap complication (flap compromise, partial and/or complete flap failure), and 4) days in hospital, defined as days in an acute in-patient hospital (i.e., not rehab or nursing facility).

DETAILED DESCRIPTION:
Infection following severe lower extremity musculoskeletal injuries is a challenging problem. Several factors hypothesized to influence infection have been explored and, in many cases, optimized or found not to be influential. A persistent area of uncertainty and variability is the timing of acute soft tissue coverage. In the United States, the mean time to coverage from injury is 10 days, and infection rates are 20-35%. In the United Kingdom, there are national guidelines to support coverage within 72 hours of injury, and infection rates are less than 10%. While the data to support early coverage is promising, the necessary evidence to make this significant change is lacking. To justify the mobilization of resources and expense required to shift practice, a definitive trial is needed. This trial seeks to fill this critical knowledge gap.

The primary objective of this trial is to determine if accelerated flap coverage (within 72 hours of injury) compared to standard flap coverage timing leads lower rates of infection and infection-related complications. The trial population includes patients 18 years and older with an acute open fracture and/or dislocation below the knee, with a diagnosed need for acute soft tissue coverage with a flap. Patients who undergo primary amputation prior to attempted flap coverage will be excluded. There will be 356 participants randomized in 1:1 ratio to receive either accelerated flap coverage (goal of flap within 72 hours from injury) or flap coverage at the time that reflects the standard of care at each institution. The timing of the trial interventions, other adjunctive treatments, the fracture fixation, and flap coverage procedures will be documented for both treatment groups. Management of the fracture or dislocation, selection of flap, and post-injury flap management will be at the discretion of the operating surgeons and documented for both treatment groups. Participants will have follow-up at 6 weeks, 3 months, 6 months, and 12 months post-randomization.

The primary outcome will be a composite outcome to evaluate clinical status 6 months after randomization. Components of the composite outcome will be hierarchically assessed in the following order: 1) all-cause mortality, 2) amputation related to injury, 3) re-operation for infection and/or flap complication (flap compromise, partial and/or complete flap failure), and 4) days in hospital, defined as days in an acute in-patient hospital (i.e., not rehab or nursing facility). The secondary outcomes will independently assess the individual components of the primary outcome at 6 and 12 months, the composite outcome at 12 months, and health-related quality of life and patient satisfaction over 6 and 12 months. An Adjudication Committee will review primary and secondary endpoints and a Data Safety Monitoring Committee (DSMC) will review all safety events.

ELIGIBILITY:
The inclusion criteria are:

1. Patients 18 years of age or older.
2. Severe lower extremity open fracture and/or dislocation below the knee requiring an acute flap for management of the musculoskeletal injury.
3. Will have all planned flap surgeries performed by a participating surgeon or delegate.
4. Able to be randomized within 48 hours of injury.

The exclusion criteria are:

1. Site is unable to implement the accelerated flap protocol due to local logistics.
2. Primary amputation anticipated prior to attempted flap for management of the injury.
3. Critical limb ischemia that requires re-vascularization for limb perfusion.
4. Chronic or acute infection at or near the musculoskeletal injury site at the time of initial injury surgery.
5. Burns at the musculoskeletal injury site.
6. Incarceration.
7. Expected injury survival of less than 12 months.
8. Terminal illness with expected survival of less than 12 months.
9. Currently enrolled in a trial that does not permit co-enrollment.
10. Declined to provide informed consent.
11. Unable to obtain informed consent due to language barriers.
12. Unable to obtain informed consent because a legally authorized representative was unavailable.
13. Anticipated problems, in the judgment of research personnel, with maintaining follow-up with the patient.
14. Prior enrollment in the trial.
15. Eligible patient or LAR was not approached within screening window (missed participant).
16. Other reason to exclude the patient, as approved by the Principal Investigators.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 356 (Estimated)
Dates: Start 2024-11-04 (Actual); Primary Completion 2029-08 (Estimated); Study Completion 2030-02 (Estimated)

PRIMARY OUTCOMES:
Clinical status | 6 months
  Clinical status is a hierarchical composite of the following outcomes:
  1. All-cause mortality
  2. Amputation related to injury
  3. Re-operation for infection and/or flap complication (flap compromise, partial and/or complete flap failure)
  4. Days in hospital, defined as days in an acute in-patient hospital (i.e., not rehab or nursing facility)

SECONDARY OUTCOMES:
Mortality | 6 months and 12 months
  All-cause mortality
Amputation | 6 months and 12 months
  Amputation related to injury. Amputation will be time-to-event, with the assumption that earlier is worse than later.
Unplanned re-operation | 6 months and 12 months
  Unplanned re-operation for infection and/or flap complication (flap compromise, partial and/or complete flap failure). Re-operation for infection and flap complication will be time-to-event, with the assumption that earlier is worse than later. Re-operation for infection and major flap complication will account for more than one operation, assuming that more operations are worse.
Number of days in hospital | 6 months and 12 months
  Days in an acute in-patient hospital (i.e., not rehab or nursing facility)
Patient-reported health status as assessed by the Euro-QoL (EQ-5D-5L) | 6 months and 12 months
  Patient-reported health status as assessed by the EQ-5D-5L. The EQ-5D-5L is scored on a 0 to 100 mm scale. 0 mm represents "the worst health you can imagine to 100 mm which represents "the best health you can imagine".
Quality of life as assessed by the Limb-Q | 6 months and 12 months
  Health-related quality of life and patient satisfaction measured with the Limb-Q. The Limb-Q is a set of independently functioning scales. All scales are scored 0-100 (higher = better). The Limb-Q Appearance, Physical, Symptoms, Financial Impact, Life Impact, and Psychological scales will be used.

CONTACTS AND LOCATIONS:
Overall Officials: Lily Mundy, MD, Principal Investigator — Johns Hopkins School of Medicine
Locations (9):
- United States (7):
  - UC Davis Medical Center, Sacramento, California
  - R Adams Cowley Shock Trauma Center, Baltimore, Maryland
  - John Hopkins Bayview Medical Center, Baltimore, Maryland
  - The Johns Hopkins Hospital, Baltimore, Maryland
  - University of Maryland Capital Region Medical Center, Largo, Maryland
  - Oregon Health & Science University, Portland, Oregon
  - Vanderbilt University Medical Center, Nashville, Tennessee
- The Alfred Hospital, Melbourne, Victoria, Australia
- Vall d'Hebron University Hospital, Barcelona, Spain